CLINICAL TRIAL: NCT06204471
Title: Evaluating the Acceptability of Airbag Hip Protectors in Older People
Brief Title: Acceptability of Hip Protector Airbags in Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Beaumont Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RFCTLR 73
Record Dates: First submitted 2023-11-14; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Falls Risk
Keywords: Hip protector; Airbag

STUDY DESIGN:
Intervention Model Description: Pilot study of two months, then crossed over to the other for two months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airbag1 (Experimental): Airbag1 worn for two months
  Interventions: Device: Helite hip protector; Device: Wolk hip protector
- Airbag2 (Experimental): Airbag2 worn for 2 months
  Interventions: Device: Helite hip protector; Device: Wolk hip protector

INTERVENTIONS:
Device: Helite hip protector — hip protector
Device: Wolk hip protector — Hip protectdor

SUMMARY:
Pilot study evaluating two different airbag hip protectors to see if community-dwelling older people will wear them and find them comfortable and acceptable.

DETAILED DESCRIPTION:
Traditional hip protectors are specialised pads designed to shield the greater trochanter on (fall) impact. They have uncertain benefits in reducing hip fracture risk and have very poor uptake due to discomfort. Recently, airbag technology has allowed radical change in design and wearability of hip protectors. Despite these airbags being commercially available, there is little evidence of their acceptability/wearability, and as with all hip protectors, virtually no research exists in community-dwelling people. A study of traditional hip protectors found that they may reduce fear of falling (FoF) in community dwellers but activity levels or quality of life were not assessed. A non-randomised study is ongoing of hip airbags on fractures in nursing homes, but none in community dwellers. Two Hip Protectors available in Europe are CE marked as personal protective equipment and approved for sale. There is a need to evaluate their acceptability and usefulness before considering larger clinical trials evaluating their efficacy in preventing hip fractures. This study will evaluate the two hip protectors and gain patient feedback in their use.

ELIGIBILITY:
Inclusion criteria:

* Age 65 years and older
* 1 or more falls in the last year requiring medical attention
* Fear of Falling (single question Y/N)
* Able to give informed consent

Exclusion criteria:

* Nursing home resident
* Immobile, or requires another person to assist with transfers and mobility
* Unable to apply or remove the hip airbag independently
* Waist circumference <70cm or >125cm (Helite device is sized by waist) and
* Hip circumference <84cm or >125cm (Wolk device sized by hip)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Acceptability and useability of a hip protector airbag, qualitative analysis | After 2 month period of wearing each airbag
  Tolerance of, and psychosocial impact of wearing a hip protector airbag will be explored through a semi-structured in-depth interview at the end of each 2-month period of wearing the airbag. This will explore significant patterns and themes related to acceptability of each airbag through deductive interview content analysis.

SECONDARY OUTCOMES:
Acceptability and useability of a hip protector airbag, quantitative measure | After 2 months of wearing each device.
  SUS (System Usability Scale): The SUS is adapted for the purposes of this study, from similar in the literature and consists of 10 questions each uses a 10 point Likert scale rating factors such as ease of use, charging the device, appearances etc. A high score (100 max score) means highly rated, and 10 (lowest score) means poorly rated.
Fear of falling (FoF) | After 2 months of wearing each device
  FoF will be assessed using the FES1 (Falls Efficacy Scale International 1) questionnaire. This uses a 4 point scale for subjective level of concern for 16 questions related to falls and activity. Maximum scores is 64 for highest level of concern or fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Dockery, MD, Principal Investigator — Beaumont Hospital
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
tbc